CLINICAL TRIAL: NCT04051502
Title: ICG-Enabled Mapping of Ovarian Sentinel Lymph Nodes: A Feasibility Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-271
Record Dates: First submitted 2019-08-05; First posted 2019-08-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer; Adnexal Mass
Keywords: Ovarian Cancer; Adnexal Mass; Ovarian Sentinal Lymph Nodes; 19-271; Memorial Sloan Kettering Cancer Center; Sentinal Lymph Nodes; indocyanine green dye; ICG Dye
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): First group of 10 participants enrolled
  Interventions: Drug: Method 1: Indocyanine green dye
- Group 2 (Experimental): Second group of 10 participants enrolled
  Interventions: Drug: Method 2: Indocyanine green dye
- Group 3 (Experimental): Third group of 10 participants enrolled
  Interventions: Drug: Method 3: Indocyanine green dye
- Group 4 (Experimental): Fourth group of 10 participants enrolled
  Interventions: Drug: Method 3: Indocyanine green dye

INTERVENTIONS:
Drug: Method 1: Indocyanine green dye — Injection 4 mL of ICG dye directly into the fallopian tube (1 or more places is acceptable) only to the side where the adnexal mass is located
  Other Names: ICG dye
  Arms: Group 1
Drug: Method 2: Indocyanine green dye — 1mL of ICG injected at each of the four sites: only to the side where the adnexal mass is located
  * Dorsal side of the IP ligament
  * Ventral side of the IP ligament
  * Dorsal side of the utero-ovarian ligament
  * Ventral side of the utero-ovarian ligament
  Other Names: ICG dye
  Arms: Group 2
Drug: Method 3: Indocyanine green dye — Injection of 2mL of ICG dye into the IP ligament pedicle after the adnexal mass has been removed. Only to the side where the adnexal mass is located
  Other Names: ICG dye
  Arms: Group 3
Drug: Method 3: Indocyanine green dye — Injection of 2mL of ICG dye into the IP ligament pedicle before the adnexal mass is removed.
  Arms: Group 4

SUMMARY:
The purpose of this study is to find out how well ovarian sentinel lymph nodes (SLNs) can be identified with indocyanine green (ICG) dye during risk-reducing ovarian surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing surgery with the Gynecology Service at MSK.
* Women undergoing surgery for an adnexal mass without pre-operative suspicion of high stage disease, with or without a hysterectomy

  °For this protocol, "suspected high stage disease" will be defined as any patient with radiologic or clinical evidence of ovarian cancer which has spread outside of the ovary. Thus, only patients with an adnexal mass, or bilateral adnexal masses, are eligible.
* Women in whom MIS surgery is converted to a laparotomy will not be excluded as both surgical approaches, MIS and open, will be utilized.
* Women >/= 18 years of age
* Able to provide informed consent
* Albumin levels within normal range

Exclusion Criteria:

* Current non-GYN primary malignancy
* Prior or current history of uterine, cervical, peritoneal, or vulvovaginal malignancy
* Ongoing anticancer therapy
* Prior bilateral oophorectomy
* Known severe anaphylactic iodide allergy
* Known history of cirrhosis or other chronic liver disease, or women with hepatic dysfunction.
* Elevated transaminases (ALT, AST) and/or Alk Phos will be evaluated by the treating physician on a case by case basis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Number and location of ovarian sentinel lymph nodes visually identified after injection of ICG dye via one of three tested methods. | 1 year
  Evaluate for dye uptake in the regional lymphatic channels, and in the pelvic and para-aortic nodes using infrared imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Ginger Gardner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only ), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org